CLINICAL TRIAL: NCT06172725
Title: Improvements by a Protein-Rich Plant-Based Diet and Resistance Exercise Program for Active Ageing
Acronym: IMPACT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amsterdam University of Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NL84531.018.23
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2023-12

CONDITIONS: Protein Intake
MeSH Terms: interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-Protein Vegetarian Diet (Experimental): High-protein vegetarian diet (no meat/fish)
  Interventions: Other: Dietary and exercise intervention
- High-Protein Omnivorous Diet (Active Comparator): High-protein omnivorous diet
  Interventions: Other: Dietary and exercise intervention

INTERVENTIONS:
Other: Dietary and exercise intervention — The healthy older adults will follow a twelve-week high-protein vegetarian diet or high-protein omnivorous diet both in combination with a resistance exercise program.
  All participants will receive blended dietary counselling. Blended dietary counselling is based on tele-coaching and face-to-face coaching performed by dieticians.

SUMMARY:
High-protein intake and physical activity are important approaches to preserve muscle mass. Consuming high levels of high-quality proteins to preserve muscle mass is challenging with a plant-based diet. The healthy, older participants will follow a twelve-week high-protein vegetarian diet or high-protein omnivorous diet both in combination with a resistance training program. The change in protein intake and muscle mass will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Aged 55 years or older
* BMI 18.5-30 kg/m2
* Living independently
* Ability and willingness to comply with the protocol
* Written an informed consent
* Consent of the study physician

Exclusion Criteria:

* Alcohol abuse (more than 14 glasses per week (women) or more than 21 glasses per week (men)) or drug abuse in the opinion of the study physician (CBS et al., 2017)
* Inability to understand the Dutch language
* Cognitive impairment (MMSE more than 25)
* Diagnosed chronic disease that may interfere with protocol (e.g., cardiovascular, gastrointestinal, neurological, known renal diseases (eGFR more than 60 mL/min (Levey & Coresh, 2012), and/or diabetes)
* Current enrolment in an exercise program or other intervention study
* Planned a holiday during the intervention period and is unable to attend training sessions for more than 1 week

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2025-06-27 (Estimated); Study Completion 2025-06-27 (Estimated)

PRIMARY OUTCOMES:
Protein intake | Three months
  Protein intake

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam University of Applied Sciences, Amsterdam, North Holland, Netherlands